CLINICAL TRIAL: NCT00536588
Title: A Phase 1 Study of the Safety and Tolerability of Intravesical Administration of SCH 721015 in Patients With Transitional Cell Carcinoma of the Bladder
Brief Title: A Safety and Tolerability Study of SCH 721015 in Patients With Transitional Cell Carcinoma of the Bladder (Study P03816)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03816
Record Dates: First submitted 2007-09-26; First posted 2007-09-28 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCH 721015 with SCH 209702 (Experimental)
  Interventions: Genetic: SCH 721015 with SCH 209702

INTERVENTIONS:
Genetic: SCH 721015 with SCH 209702 — Each subject receives a single intravesical administration of SCH 721015 with SCH 209702 at dose levels of 1 x 10^9 to 3 x 10^11 particles/mL (based on assessment of tolerability, intermediate dose levels may be used).

SUMMARY:
The purpose of this first-in-human study is to determine the safety and tolerability of SCH 721015 in subjects with transitional cell carcinoma of the bladder.

DETAILED DESCRIPTION:
A nonrandomized, open-label, rising-dose, parallel-group, multi-center study of SCH 721015 in patients with papillary bladder cancer, or carcinoma in situ that is refractory to Bacillus Calmette-Guerin. Subjects will receive a single intravesical administration of SCH 721015 with SCH 209702 in a total volume of 75 mL with a 1-hour dwell time. Subjects who at 3 months post administration demonstrate a complete response (CR on cystoscopy/biopsy and cytology) and who did not experience dose-limiting toxicity will be allowed to receive a second intravesical administration at the same dose level.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven recurrent transitional cell carcinoma of the bladder, Stage Tis, Ta.
* Patients with recurrent T1 disease who do not wish to have cystectomy.
* Subjects must have failed at least two prior courses of BCG with or without recombinant interferon alpha administration.
* At least 3 months must have passed since last intravesical treatment for bladder carcinoma.
* Subjects must be 18 years of age or older.
* Life expectancy of at least 3 months.
* Adequate performance status (Karnofsky score >=70%).
* Adequate laboratory values.

Exclusion Criteria:

* Suspected hypersensitivity to interferon alpha.
* Subjects with organ transplants.
* Any known preexisting medical condition that could interfere with the subject's participation in and completion of the study such as:

  * History of psychosis or presence of poorly controlled depression;
  * CNS trauma or active seizure disorders requiring medication;
  * Significant cardiovascular dysfunction within the past 6 months including symptomatic cardiac ischemia, arrhythmia or congestive heart failure requiring hospitalization or emergency room visit within last 3 months;
  * Poorly controlled diabetes mellitus (HbA1C >10.0%);
  * Unstable chronic pulmonary disease requiring hospitalization or emergency room visit within the last 3 months;
  * Immunologically mediated disease (eg, rheumatoid arthritis, autoimmune hepatitis, immune mediated glomerulonephritis).
* History of any clinically significant local or systemic infectious disease within 4 weeks prior to initial treatment administration.
* Untreated bladder infection.
* Positive for hepatitis BsAg or HIV Ab or hepatitis C.
* Immunosuppressive therapy within the last 3 months.
* BCG therapy or intravesical therapy within 3 months.
* Traumatic catheterization within 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Adverse events, laboratory safety tests, dose-limiting toxicity | CBC/chemistry: predose, Days 1-3, 7, 14, 21, & 28, Week 12.
Adverse events, laboratory safety tests, dose-limiting toxicity | Additional hematology on Days 4, 5, & 6.
Adverse events, laboratory safety tests, dose-limiting toxicity | AEs: Duration of study; up to 3 years postdose for serious events.
Adverse events, laboratory safety tests, dose-limiting toxicity | ECG and VS - predose and selected postdose time points.

SECONDARY OUTCOMES:
Timed urine collections for IFNα2b excretion & IP-10. | Days 1-7, 10, 14, 21, & 28/29.
Urine samples for SCH 721015 DNA content. | Predose, Days 1-7 & 14.
Blood samples for SCH 721015 DNA; SCH 209702, & IFNα2b levels; antiadenoviral & anti-IFNα2b antibodies | Pre- & postdose for SCH 721015 DNA; SCH 721015, & IFNα2b levels; & postdose for antibodies.
Urine cytology & FISH | Days 1, 30 & 90
Cystoscopy & bladder biopsies | Screening & Day 90

REFERENCES:
- [Result] Dinney CP, Fisher MB, Navai N, O'Donnell MA, Cutler D, Abraham A, Young S, Hutchins B, Caceres M, Kishnani N, Sode G, Cullen C, Zhang G, Grossman HB, Kamat AM, Gonzales M, Kincaid M, Ainslie N, Maneval DC, Wszolek MF, Benedict WF. Phase I trial of intravesical recombinant adenovirus mediated interferon-alpha2b formulated in Syn3 for Bacillus Calmette-Guerin failures in nonmuscle invasive bladder cancer. J Urol. 2013 Sep;190(3):850-6. doi: 10.1016/j.juro.2013.03.030. Epub 2013 Mar 15. PMID 23507396